CLINICAL TRIAL: NCT00002558
Title: PHASE I/II TRIAL OF SEQUENTIAL TAXOL/IFOSFAMIDE AND DOSEINTENSIVE CARBOPLATIN/ETOPOSIDE WITH STEM CELL SUPPORT IN CISPLATIN-RESISTANT GERM CELL TUMOR PATIENTS WITH UNFAVORABLE PROGNOSTIC FEATURES
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Germ Cell Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 93-162; P30CA008748 (NIH); MSKCC-93162; NCI-V94-0407
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Extragonadal Germ Cell Tumor; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: recurrent malignant testicular germ cell tumor; recurrent ovarian germ cell tumor; extragonadal germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Filgrastim; Carboplatin; Etoposide; Ifosfamide; Paclitaxel; Peripheral Blood Stem Cell Transplantation

ARMS (1):
- chemotherapy administered with G-CSF and PBSC support (Experimental): The design of this trial is a phase I/II trial of sequential accelerated chemotherapy cycles with taxol/ifosfamide and carboplatin/etoposide administered with G-CSF and PBSC support.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: etoposide; Drug: ifosfamide; Drug: paclitaxel; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: etoposide
Drug: ifosfamide
Drug: paclitaxel
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, ifosfamide, carboplatin, and etoposide work in different ways to stop the growth of tumor cells, either by killing them or by stopping them from dividing. Giving chemotherapy with a peripheral stem cell transplant may allow more chemotherapy to be given so that more tumor cells are killed.

The design of this trial is a phase I/II trial of sequential accelerated chemotherapy cycles with taxol/ifosfamide and carboplatin/etoposide administered with G-CSF and PBSC support.

PURPOSE: The purpose of this study is to determine the effects of an intensive sequence of chemotherapy drugs in patients with metastatic germ cell cancer. All of these chemotherapy drugs are known to be active in this disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of paclitaxel and ifosfamide followed by carboplatin and etoposide with stem cell support in patients with unfavorable germ cell tumors with unfavorable prognostic factors and resistance to cisplatin.
* Determine the efficacy of this regimen as salvage therapy in these patients.
* Escalate the dose of carboplatin based on a target area under the concentration time curve and renal function, and determine the pharmacokinetics of carboplatin in selected patients.
* Determine the qualitative effects of paclitaxel and ifosfamide on hematopoietic progenitors in these patients.

OUTLINE: This is a dose escalation study of carboplatin.

* Part A: Patients receive paclitaxel IV continuously on day 1 and ifosfamide IV over 4 hours on days 2-4. Autologous peripheral blood stem cells (PBSC) are harvested on days 11-13. Filgrastim (G-CSF) is administered subcutaneously (SC) twice daily beginning 6 hours after completion of paclitaxel and ifosfamide infusions and continuing until the last day of leukapheresis. Treatment continues every 2 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Before beginning the first course of chemotherapy, autologous bone marrow (ABM) is harvested, if possible, in case insufficient peripheral blood stem cells (PBSC) are harvested. Patients who were unable to undergo harvest of ABM before the first course of chemotherapy undergo harvest of ABM before beginning the second course of chemotherapy.
* Part B : Beginning 2 weeks after completion of regimen A, patients receive etoposide IV over 2 hours and carboplatin IV over 1 hour on days 1-3. PBSC are reinfused on day 5. G-CSF is administered SC twice daily beginning 6 hours after completion of etoposide and carboplatin infusions and continuing until blood counts recover. G-CSF is held on the morning of PBSC transplantation and restarted beginning 6 hours after completion of PBSC transplantation. Treatment continues every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients with insufficient PBSC for the second course receive PBSC combined with ABM. Patients with insufficient PBSC for the third course receive ABM.

During the second part, cohorts of 3-6 patients receive escalating doses of carboplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose-limiting toxicity.

After completion of parts A and B, some patients may undergo resection of residual masses.

ELIGIBILITY:
Inclusion criteria:

* Male/Female with histologically confirmed GCT with review by the Department of Pathology at this center.
* Patients with advanced GCT, including patients with:

measurable or evaluable disease,

* patients with only elevated serum tumor markers (AFP and/or HCG), or
* patients with known residual disease after postchemotherapy surgery. Eligible patients must have established clinical resistance to cisplatin by their failure to achieve a durable CR to a cisplatin-based regimen.
* Prior treatment limited to ≤ 6 prior cycles (≤ four cycles preferred) of cisplatin. (GROUP A)
* Prior therapy > 6 cycles of cisplatin. (GROUP B)
* Therapy must have been discontinued at least 3 weeks before entry onto protocol.
* Patients must have one or more unfavorable prognostic factors for achieving a CR to cisplatin-based salvage therapy. These are:
* Extragonadal primary site.
* Testis/ovarian primary site with the best response of an IR to first-line therapy, or a partial response with normal tumor markers of six months or less in duration.
* Prior treatment with ifosfamide-containing therapy
* General medical condition sufficient to allow for general anesthesia at the time of pheresis catheter placement.
* Patients must have negative serology for Human Immunodeficiency Virus.
* Laboratory criteria for protocol entry:

WBC ≥ 3000/ul Platelets 3 100,000/ul Cr Clearance > 50 cc/min*

* (unless renal dysfunction is due to tumor obstructing the ureters in which case eligibility will be determined by the Principal Investigator).

* Age ≥ 15 years.
* Signed informed consent.

Exclusion Criteria:

* Presence of active infection
* Concurrent treatment with chemotherapy or
* Inability to comply with the treatment protocol or to undergo the specified follow-up tests for safety or effectiveness.
* Prior high-dose therapy with AuBMT.
* Patients must have recovered from recent surgery.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 1994-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gnanamba V. Kondagunta, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Feldman DR, Sheinfeld J, Bajorin DF, Fischer P, Turkula S, Ishill N, Patil S, Bains M, Reich LM, Bosl GJ, Motzer RJ. TI-CE high-dose chemotherapy for patients with previously treated germ cell tumors: results and prognostic factor analysis. J Clin Oncol. 2010 Apr 1;28(10):1706-13. doi: 10.1200/JCO.2009.25.1561. Epub 2010 Mar 1. PMID 20194867
- [Result] Kondagunta GV, Bacik J, Sheinfeld J, Bajorin D, Bains M, Reich L, Deluca J, Budnick A, Ishill N, Mazumdar M, Bosl GJ, Motzer RJ. Paclitaxel plus Ifosfamide followed by high-dose carboplatin plus etoposide in previously treated germ cell tumors. J Clin Oncol. 2007 Jan 1;25(1):85-90. doi: 10.1200/JCO.2006.06.9401. PMID 17194908

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Group A: Prior Treatment Limited to <= 6 Cycles of Cisplatin
- Group B: Group B: Prior Treatment Limited to > 6 Cycles of Cisplatin
Period: Overall Study
Arm/Group | Group A | Group B
Started | 92 | 16
Completed | 92 | 15
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 92 | 16 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3
  Between 18 and 65 years | 89 | 16 | 105
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 90 | 15 | 105

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Overall Objective Response will be assessed prior to dose-intensive therapy and at the completion of therapy. Complete disappearance of all clinical, radiographic and biochemical (normal AFP and HCG) evidence of disease for a minimum of 4 weeks (CR to chemotherapy). Patients must be free of disease for a minimum of 4 weeks. Partial Response: Complete disappearance of all biochemical evidence of disease in patients without a surgical procedure for a residual radiographic mass. Patients must demonstrate no biochemical recurrence or progression of radiographic masses for a minimum of four weeks (PR to chemotherapy}
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 91 | 15
participants
  Complete Response (CR) | 50 | 4
  Incomplete Response (IR) | 36 | 8
  Partial Response (PR) | 5 | 3

ADVERSE EVENTS:
Groups:
- Group A: <= 6 Cycles of Cisplatin: Group A: Prior Treatment Limited to <= 6 Cycles of Cisplatin
- Group: B > 6 Cycles of Cisplatin: Group B: Prior Treatment Limited to > 6 Cycles of Cisplatin
Arm/Group | Group A: <= 6 Cycles of Cisplatin | Group: B > 6 Cycles of Cisplatin
Serious Adverse Events (participants affected / at risk) | 7/92 | 2/16
Other Adverse Events (participants affected / at risk) | 92/92 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: <= 6 Cycles of Cisplatin (N=92) | Group: B > 6 Cycles of Cisplatin (N=16)
CNS hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (General disorders) | 1 (1) | 0 (0)
Neurology, other (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Syncope (General disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: <= 6 Cycles of Cisplatin (N=92) | Group: B > 6 Cycles of Cisplatin (N=16)
Abdominal pain/cramping (Gastrointestinal disorders) | 8 (8) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 16 (16) | 3 (3)
Alopecia (General disorders) | 0 (0) | 1 (1)
Bilirubin (Metabolism and nutrition disorders) | 23 (23) | 4 (4)
Catheter-related infection (Infections and infestations) | 6 (6) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 8 (8) | 3 (3)
Dermatology, skin other (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Edema (General disorders) | 0 (0) | 1 (1)
Erythema multiforme (Cardiac disorders) | 5 (5) | 0 (0)
Fatigue (General disorders) | 22 (22) | 2 (2)
Fever (General disorders) | 26 (26) | 4 (4)
Hearing, other (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 92 (92) | 15 (15)
Hemorrhage, other (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 80 (80) | 12 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 12 (12) | 0 (0)
Hypermagnesmia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (12) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 51 (51) | 11 (11)
Hypoglycemia (Metabolism and nutrition disorders) | 19 (19) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 44 (44) | 8 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 65 (65) | 10 (10)
Hyponatremia (Metabolism and nutrition disorders) | 30 (30) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 63 (63) | 13 (13)
Hypotension (Cardiac disorders) | 6 (6) | 2 (2)
Infection with grade 3/4 neutopenia (Infections and infestations) | 5 (5) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 90 (90) | 15 (15)
Lymphopenia (Blood and lymphatic system disorders) | 91 (91) | 15 (15)
Neuropathy-sensory (Nervous system disorders) | 0 (0) | 2 (2)
Neutrophils (Blood and lymphatic system disorders) | 89 (89) | 15 (15)
Pain, other (General disorders) | 7 (7) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 89 (89) | 15 (15)
Prothrombin time (PT) (Blood and lymphatic system disorders) | 16 (16) | 1 (1)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 10 (10) | 3 (3)
Rash, desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SGOT (AST) (Blood and lymphatic system disorders) | 17 (17) | 0 (0)
SGPT (ALT) (Blood and lymphatic system disorders) | 24 (24) | 2 (2)
Thrombosis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (10) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes